CLINICAL TRIAL: NCT06339255
Title: A Multicenter Prospective Observational Study on Chimeric Antigen Receptor (CAR) T-cell Therapy for Lymphoma: Monitoring Feasibility, Efficacy, Toxicity and Biomarkers in a Real Life Setting
Brief Title: Italian Observational Study on CAR-T Therapy for Lymphoma
Acronym: CART-SIE
Status: Recruiting | Type: Observational
Sponsor: Paolo Corradini (Other)
Collaborators: Annalisa Chiappella (Unknown); Cristiana Carniti (Unknown); Anna Dodero (Unknown)
Responsible Party: Sponsor-Investigator, Paolo Corradini, Professor, director of hematology Unit, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Organization: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Other Study IDs: INT 180/19
Record Dates: First submitted 2024-01-04; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Diffuse Low Grade B-Cell Lymphoma; Primary Mediastinal Large B-cell Lymphoma (PMBCL); Mantle Cell Lymphoma; Follicular Lymphoma
Keywords: CAR-T; Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Diagnostic tissue block or 10 unstained slides to be collected at study entry. Fresh LK product for immune monitoring. Perifheral blood samples collected at defined timepoints, from screeining to follow-up phase, until relapse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study on chimeric antigen receptor T-cell therapy is to monitor the feasibility, efficacy, toxicity and biomarkers in a real life setting.

Partecipants will be asked to agree to their clinical data collection and to partecipate to the optional biological study that aims to evaluate biomarkers of toxicity and response (clinical characteristics, cytokine profile, cellcomposition and type of the CAR-T cell product, lymphoma genomics). The study will evaluate even the disease response according to lugano criteria by PET and CT in routine clinical activity.

DETAILED DESCRIPTION:
This observational prosopective multicenter study aims to:

1. evaluate the feasibility of CAR T-cell treatment in the real-life setting, with particular regard to eligible patients versus those subjected to leukapheresis versus those finally treated.
2. evaluate the survival outcome of PMBCL, DLBCL, MCL and FL patients treated with CAR T-cells versus those potentially eligible, but excluded from cellular therapy for other causes (either related to the patient or to the manufacturing);
3. monitor the incidence of early and late AEs up to three year after CAR-T;
4. evaluate disease response and immune recovery biomarkers at different time-points up after CAR-T (when clinically indicated or using blood sampling leftover);
5. evaluate biomarkers of toxicity and response (clinical characteristics, cytokine profile, cell composition and type of the CAR T-cell product, lymphoma genomics).
6. evaluate disease response according to Lugano criteria by PET and CT in routine clinical activity.

Primary Objective:

• Feasibility and efficacy of the treatment in the real life practice

Secondary Objectives:

* Evaluation of Outcome [Response rate (ORR), Overall survival (OS), Progression free survival (PFS), duration of response (DoR) non-relapse mortality (NRM)] according to Lugano criteria.
* Evaluation of safety (CRS, neurotoxicity, infections, cytopenias, B cell aplasia, second malignancies) with particular attention to the safety in the new indications
* Evaluation of bridging therapy (outcome and safety)
* Evaluation of salvage therapy after CAR-T failure (outcome and safety)
* Comparison of the different CAR T-cell products (time from patient screening to infusion, disease response and safety)
* Comparison of the different histotypes (PMBCL, DLBCL, MCL FL) according to CAR-T cell products

Biological Studies

* Characterization of biomarkers of early response (circulating tumor cell free DNA versus PET and CT scans)
* Characterization of toxicity biomarkers
* Analysis of the immune reconstitution and CAR-T expression Radiomics Evaluation
* Influence of PET quantitative parameters (tMTV, Distance max, Distance max bulky, metabolic changes between baseline and +30 and +90 after CAR T-cell infusion (ΔSUV max) on outcome
* Influence of PET quantitative parameters (tMTV, Distance max, Distance max bulky, metabolic changes between baseline and +30 and +90 after CAR T-cell infusion (ΔSUV max) on outcome.

Primary endpoint:

to evaluate the percentage of patients infused versus those eligible and leukoapheresed to evaluate the overall response and survival at one year of the patients treated with CAR T cells.

Secondary endpoints:

Overall response rate (ORR) at 3-6-12-18 months Overall survival (OS) for all patients included in the study OS, Progression free survival (PFS), Event free survival (EFS), and duration of response (DoR), non-relapse mortality (NRM) after CAR T-cell therapy at one,two years and 5 years Incidence and grading of CRS and neurotoxicity Number of patients receiving a bridging therapy before lymphodepletion Intensive Care Unit admission rate for all treated patients Lymphoma genomics and circulating cell free DNA as early response biomarker Characterization of toxicity biomarkers Analysis of immune reconstitution and CAR-T expression Early Adverse event (grading/onset/severity/treatment) Long term Safety (AE grading/onset/severity/treatment) Incidence of second malignancies Evaluation of quantitative parameters of PET by central review, when applicable in selected sites This is an observational multicenter prospective study enrolling all consecutive patients referred to the Italian hematologic centers already qualified for CAR T-cell treatment with relapsed/refractory DLBCL, PMBCL, MCL and FL. The screening will be done according to the axi-cel, tisagen-cel, brexucabtagene autoleucel and lisocabtagene maraleucel label criteria, the eligibility of a given patient to CAR-T will be definedaccording to AIFA criteria.

All patients eligible to CAR-T will be consecutively enrolled Biological samples will be stored at each institution or centralized at the Fondazione IRCCS Istituto Nazionale dei Tumori, Milano. Fondazione Italiana Linfomi (FIL) will be in charge of the GCP management of the study. Web-based CRF are prepared by FIL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of DLCBL, PMBCL, MCL and FL eligible for CAR-T treatment with commercialy available products in Italy.

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of DLCBL, PMBCL, MCL and FL eligible for CAR-T treatment with commercialy available products in Italy.
Sampling Method: Probability Sample
Enrollment: 5300 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the CAR-T cells treatment in lymphomas in the italian real life practice | 10 years enrollment, minimum 1 year follow-up
  Evaluate the feasibility of CAR T-cell treatment in the real-life setting, with particular regard to eligible patients versus those subjected to leukapheresis versus those finally treated. The percentage of patients infused will be estimated as the number of patients infused divided by the total number of those declared eligible; the corresponding exact confidence intervals at 95% will also be estimated.
Efficacy of the CAR-T cells treatment in lymphomas in the italian real life practice | 10 years enrollment, minimum 1 year follow-up
  Evaluate the survival outcome of PMBCL, DLBCL, MCL and FL patients treated with CAR T-cells versus those potentially eligible, but excluded from cellular therapy for other causes (either related to the patient or to the manufacturing)

SECONDARY OUTCOMES:
Evaluation of Outcome: Overall Response rate (ORR), according to Lugano criteria. | 10 years, minimum f-up 1 year
  Overall response rate (ORR): the percentage of responding patients will be estimated as the number of patients with complete response (CR) + partial response (PR) divided by the total number of patients assessable at each specific timepoint (3-6-12-18 months). Patients not assessable for response for any reason will be considered as non-responding in the calculation of the response rate. The exact 95% confidence intervals of the response percentage will also be estimated.
Evaluation of Outcome: Overall survival (OS), according to Lugano criteria. | 10 years, minimum f-up 1 year
  Overall survival (OS): time will be measured as the interval between the date of CAR-T infusion and the date of death for all causes, with censoring at the date of the latest follow-up in alive patients. OS curves will be estimated with the Kaplan Meier method.
Evaluation of Outcome: Progression free survival (PFS) | 10 years, minimum f-up 1 year
  Progression-free survival (PFS): time will be measured as the interval between the CAR-T infusion and the date of progression disease (PD), or death, whichever occurs first.
Evaluation of Outcome: duration of response (DoR) | 10 years, minimum f-up 1 year
  Duration of Response (DoR): for patients who will respond to treatment, the duration of response will be measured as the interval between the response achievement and the date of progression or death, whichever occurs first, with censoring at the date of the latest follow-up in alive patients without progression. DoR curves will be estimated with the Kaplan Meier method.
Evaluation of Outcome: Overall Response rate (ORR) | 10 years, minimum f-up 1 year
  Overall response rate (ORR): the percentage of responding patients will be estimated as the number of patients with complete response (CR) + partial response (PR) divided by the total number of patients assessable at each specific timepoint (3-6-12-18 months). Patients not assessable for response for any reason will be considered as non-responding in the calculation of the response rate. The exact 95% confidence intervals of the response percentage will also be estimated.
Evaluation of Outcome: Overall survival (OS) | 10 years, minimum f-up 1 year
  Overall survival (OS): time will be measured as the interval between the date of CAR-T infusion and the date of death for all causes, with censoring at the date of the latest follow-up in alive patients. OS curves will be estimated with the Kaplan Meier method.
Evaluation of Outcome: non-relapse mortality (NRM) | 10 years, minimum f-up 1 year
  Non-relapse mortality (NRM) after CAR-T cell therapy: time will be measured as the interval between the date of treatment start and the date of non-relapse death, with censoring at the date of the latest follow-up in alive patients without relapse. NRM cumulative incidence curves will be estimated regarding disease recurrence as competing event, and between groups comparisons will be performed using the Gray test.
Evaluation of safety (CRS, neurotoxicity, infections, cytopenias, B cell aplasia, second malignancies) with particular attention to the safety in the new indications | 10 years, minimum f-up 1 year
  CRS and ICANS will be measured according to ASCTC. Other toxicities will be measured according to CTCAE.
Evaluation of bridging therapy: safety | 10 years, minimum f-up 1 year
  Bridging therapy will be analysed in terms of safety as per adverse event occurrence (according to CTCAE).
Evaluation of bridging therapy: efficay | 10 years, minimum f-up 1 year
  Bridging therapy will be analysed in terms of efficacy in terms of response achievement compared to response assessment prior to bridging therapy.
Evaluation of salvage therapy after CAR-T failure | 10 years, minimum f-up 1 year
  In case of relapse after CAR-T, data regarding salvage therapy will be collected in terms of reponse (PFS)
Evaluation of salvage therapy after CAR-T failure | 10 years, minimum f-up 1 year
  In case of relapse after CAR-T, data regarding salvage therapy will be collected in terms of survival (OS).
Comparison of the different CAR T-cell products (time from patient screening to infusion, disease response and safety) | 10 years, minimum f-up 1 year
  Time form screening to infusion will be compared between CAR-T products, disease response will be evaluated in terms of CR, PR and SD.
Comparison of the different histotypes (PMBCL, DLBCL, MCL FL) according to CAR-T cell products | 10 years, minimum f-up 1 year
  Study popoulation will be analysed in terms of reponse and type CAR-T product.

OTHER OUTCOMES:
Characterization of biomarkers of early response (circulating tumor cell free DNA versus PET and CT scans) | 10 years, minimum f-up 1 year
  To study the circulating cell free DNA modulation during time, besides descriptive statistical analyses, we will use non parametric factorial models for longitudinal data [Brunner E, Domhof S, Langer F. Nonparametric analysis of longitudinal data in factorial experiments. John Wiley & Sons 2002, New York]. Such models were chosen because they allow take into account measurement incompleteness and positive asymmetry of biomarker distribution, and because they are robust to outliers. The models also allow to test the difference in the longitudinal profiles according to specific covariates.
Characterization of toxicity biomarkers | 10 years, minimum f-up 1 year
  Biomarkers will be analysed in relation to toxicities occurrence on order to identify predictors of toxicity onset and severity
Analysis of the immune reconstitution | 10 years, minimum f-up 1 year
  Evaluate disease response and immune recovery biomarkers at different time-points up after CAR-T (when clinically indicated or using blood sampling leftover)
Analysis of the CAR-T expression | 10 years, minimum f-up 1 year
  Evaluate the persistence of CAR-T after administration
Influence of PET quantitative parameters: tMTV changes between baseline and +30 and +90 after CAR T-cell infusion (ΔSUV max) related to outcome | 10 years, minimum f-up 1 year
  In our study, the PET scans will be collected and anonymized. A central review with analyses of quantitative parameters will be performed. Evaluation of baseline tMTV calculated by MTV4 method which automatically segments area with SUV ≥4.0.
Influence of PET quantitative parameters: Distance max | 10 years, minimum f-up 1 year
  In our study, the PET scans will be collected and anonymized. A central review with analyses of quantitative parameters will be performed. Dmax between baseline and +30 and +90 after CAR-T cells infusion
Influence of PET quantitative parameters: Distance max bulky | 10 years, minimum f-up 1 year
  In our study, the PET scans will be collected and anonymized. A central review with analyses of quantitative parameters will be performed. Dmax bulk is the maximum distance to the bulk and we wil analyse its change between baseline and day +30 and +90.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crump M, Neelapu SS, Farooq U, Van Den Neste E, Kuruvilla J, Westin J, Link BK, Hay A, Cerhan JR, Zhu L, Boussetta S, Feng L, Maurer MJ, Navale L, Wiezorek J, Go WY, Gisselbrecht C. Outcomes in refractory diffuse large B-cell lymphoma: results from the international SCHOLAR-1 study. Blood. 2017 Oct 19;130(16):1800-1808. doi: 10.1182/blood-2017-03-769620. Epub 2017 Aug 3. PMID 28774879
- [Result] Neelapu SS, Locke FL, Bartlett NL, Lekakis LJ, Miklos DB, Jacobson CA, Braunschweig I, Oluwole OO, Siddiqi T, Lin Y, Timmerman JM, Stiff PJ, Friedberg JW, Flinn IW, Goy A, Hill BT, Smith MR, Deol A, Farooq U, McSweeney P, Munoz J, Avivi I, Castro JE, Westin JR, Chavez JC, Ghobadi A, Komanduri KV, Levy R, Jacobsen ED, Witzig TE, Reagan P, Bot A, Rossi J, Navale L, Jiang Y, Aycock J, Elias M, Chang D, Wiezorek J, Go WY. Axicabtagene Ciloleucel CAR T-Cell Therapy in Refractory Large B-Cell Lymphoma. N Engl J Med. 2017 Dec 28;377(26):2531-2544. doi: 10.1056/NEJMoa1707447. Epub 2017 Dec 10. PMID 29226797
- [Result] Locke FL, Ghobadi A, Jacobson CA, Miklos DB, Lekakis LJ, Oluwole OO, Lin Y, Braunschweig I, Hill BT, Timmerman JM, Deol A, Reagan PM, Stiff P, Flinn IW, Farooq U, Goy A, McSweeney PA, Munoz J, Siddiqi T, Chavez JC, Herrera AF, Bartlett NL, Wiezorek JS, Navale L, Xue A, Jiang Y, Bot A, Rossi JM, Kim JJ, Go WY, Neelapu SS. Long-term safety and activity of axicabtagene ciloleucel in refractory large B-cell lymphoma (ZUMA-1): a single-arm, multicentre, phase 1-2 trial. Lancet Oncol. 2019 Jan;20(1):31-42. doi: 10.1016/S1470-2045(18)30864-7. Epub 2018 Dec 2. PMID 30518502
- [Result] Neelapu SS, Jacobson CA, Ghobadi A, Miklos DB, Lekakis LJ, Oluwole OO, Lin Y, Braunschweig I, Hill BT, Timmerman JM, Deol A, Reagan PM, Stiff P, Flinn IW, Farooq U, Goy AH, McSweeney PA, Munoz J, Siddiqi T, Chavez JC, Herrera AF, Bartlett NL, Bot AA, Shen RR, Dong J, Singh K, Miao H, Kim JJ, Zheng Y, Locke FL. Five-year follow-up of ZUMA-1 supports the curative potential of axicabtagene ciloleucel in refractory large B-cell lymphoma. Blood. 2023 May 11;141(19):2307-2315. doi: 10.1182/blood.2022018893. PMID 36821768
- [Result] Schuster SJ, Tam CS, Borchmann P, Worel N, McGuirk JP, Holte H, Waller EK, Jaglowski S, Bishop MR, Damon LE, Foley SR, Westin JR, Fleury I, Ho PJ, Mielke S, Teshima T, Janakiram M, Hsu JM, Izutsu K, Kersten MJ, Ghosh M, Wagner-Johnston N, Kato K, Corradini P, Martinez-Prieto M, Han X, Tiwari R, Salles G, Maziarz RT. Long-term clinical outcomes of tisagenlecleucel in patients with relapsed or refractory aggressive B-cell lymphomas (JULIET): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2021 Oct;22(10):1403-1415. doi: 10.1016/S1470-2045(21)00375-2. Epub 2021 Sep 10. PMID 34516954
- [Result] Abramson JS, Palomba ML, Gordon LI, Lunning MA, Wang M, Arnason J, Mehta A, Purev E, Maloney DG, Andreadis C, Sehgal A, Solomon SR, Ghosh N, Albertson TM, Garcia J, Kostic A, Mallaney M, Ogasawara K, Newhall K, Kim Y, Li D, Siddiqi T. Lisocabtagene maraleucel for patients with relapsed or refractory large B-cell lymphomas (TRANSCEND NHL 001): a multicentre seamless design study. Lancet. 2020 Sep 19;396(10254):839-852. doi: 10.1016/S0140-6736(20)31366-0. Epub 2020 Sep 1. PMID 32888407
- [Result] Locke FL, Miklos DB, Jacobson CA, Perales MA, Kersten MJ, Oluwole OO, Ghobadi A, Rapoport AP, McGuirk J, Pagel JM, Munoz J, Farooq U, van Meerten T, Reagan PM, Sureda A, Flinn IW, Vandenberghe P, Song KW, Dickinson M, Minnema MC, Riedell PA, Leslie LA, Chaganti S, Yang Y, Filosto S, Shah J, Schupp M, To C, Cheng P, Gordon LI, Westin JR; All ZUMA-7 Investigators and Contributing Kite Members. Axicabtagene Ciloleucel as Second-Line Therapy for Large B-Cell Lymphoma. N Engl J Med. 2022 Feb 17;386(7):640-654. doi: 10.1056/NEJMoa2116133. Epub 2021 Dec 11. PMID 34891224
- [Result] Abramson JS, Solomon SR, Arnason J, Johnston PB, Glass B, Bachanova V, Ibrahimi S, Mielke S, Mutsaers P, Hernandez-Ilizaliturri F, Izutsu K, Morschhauser F, Lunning M, Crotta A, Montheard S, Previtali A, Ogasawara K, Kamdar M. Lisocabtagene maraleucel as second-line therapy for large B-cell lymphoma: primary analysis of the phase 3 TRANSFORM study. Blood. 2023 Apr 6;141(14):1675-1684. doi: 10.1182/blood.2022018730. PMID 36542826
- [Result] Wang M, Munoz J, Goy A, Locke FL, Jacobson CA, Hill BT, Timmerman JM, Holmes H, Jaglowski S, Flinn IW, McSweeney PA, Miklos DB, Pagel JM, Kersten MJ, Milpied N, Fung H, Topp MS, Houot R, Beitinjaneh A, Peng W, Zheng L, Rossi JM, Jain RK, Rao AV, Reagan PM. KTE-X19 CAR T-Cell Therapy in Relapsed or Refractory Mantle-Cell Lymphoma. N Engl J Med. 2020 Apr 2;382(14):1331-1342. doi: 10.1056/NEJMoa1914347. PMID 32242358
- [Result] Monfrini C, Stella F, Aragona V, Magni M, Ljevar S, Vella C, Fardella E, Chiappella A, Nanetti F, Pennisi M, Dodero A, Guidetti A, Corradini P, Carniti C. Phenotypic Composition of Commercial Anti-CD19 CAR T Cells Affects In Vivo Expansion and Disease Response in Patients with Large B-cell Lymphoma. Clin Cancer Res. 2022 Aug 2;28(15):3378-3386. doi: 10.1158/1078-0432.CCR-22-0164. PMID 35583610
- [Result] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Result] Biancon G, Gimondi S, Vendramin A, Carniti C, Corradini P. Noninvasive Molecular Monitoring in Multiple Myeloma Patients Using Cell-Free Tumor DNA: A Pilot Study. J Mol Diagn. 2018 Nov;20(6):859-870. doi: 10.1016/j.jmoldx.2018.07.006. Epub 2018 Aug 28. PMID 30165206
- [Result] Chapuy B, Stewart C, Dunford AJ, Kim J, Kamburov A, Redd RA, Lawrence MS, Roemer MGM, Li AJ, Ziepert M, Staiger AM, Wala JA, Ducar MD, Leshchiner I, Rheinbay E, Taylor-Weiner A, Coughlin CA, Hess JM, Pedamallu CS, Livitz D, Rosebrock D, Rosenberg M, Tracy AA, Horn H, van Hummelen P, Feldman AL, Link BK, Novak AJ, Cerhan JR, Habermann TM, Siebert R, Rosenwald A, Thorner AR, Meyerson ML, Golub TR, Beroukhim R, Wulf GG, Ott G, Rodig SJ, Monti S, Neuberg DS, Loeffler M, Pfreundschuh M, Trumper L, Getz G, Shipp MA. Molecular subtypes of diffuse large B cell lymphoma are associated with distinct pathogenic mechanisms and outcomes. Nat Med. 2018 May;24(5):679-690. doi: 10.1038/s41591-018-0016-8. Epub 2018 Apr 30. PMID 29713087
- [Result] Orlando EJ, Han X, Tribouley C, Wood PA, Leary RJ, Riester M, Levine JE, Qayed M, Grupp SA, Boyer M, De Moerloose B, Nemecek ER, Bittencourt H, Hiramatsu H, Buechner J, Davies SM, Verneris MR, Nguyen K, Brogdon JL, Bitter H, Morrissey M, Pierog P, Pantano S, Engelman JA, Winckler W. Genetic mechanisms of target antigen loss in CAR19 therapy of acute lymphoblastic leukemia. Nat Med. 2018 Oct;24(10):1504-1506. doi: 10.1038/s41591-018-0146-z. Epub 2018 Oct 1. PMID 30275569
- [Result] Singh N, Perazzelli J, Grupp SA, Barrett DM. Early memory phenotypes drive T cell proliferation in patients with pediatric malignancies. Sci Transl Med. 2016 Jan 6;8(320):320ra3. doi: 10.1126/scitranslmed.aad5222. PMID 26738796
- [Result] Hirayama AV, Gauthier J, Hay KA, Voutsinas JM, Wu Q, Gooley T, Li D, Cherian S, Chen X, Pender BS, Hawkins RM, Vakil A, Steinmetz RN, Acharya UH, Cassaday RD, Chapuis AG, Dhawale TM, Hendrie PC, Kiem HP, Lynch RC, Ramos J, Shadman M, Till BG, Riddell SR, Maloney DG, Turtle CJ. The response to lymphodepletion impacts PFS in patients with aggressive non-Hodgkin lymphoma treated with CD19 CAR T cells. Blood. 2019 Apr 25;133(17):1876-1887. doi: 10.1182/blood-2018-11-887067. Epub 2019 Feb 19. PMID 30782611
- [Result] Kochenderfer JN, Somerville RPT, Lu T, Shi V, Bot A, Rossi J, Xue A, Goff SL, Yang JC, Sherry RM, Klebanoff CA, Kammula US, Sherman M, Perez A, Yuan CM, Feldman T, Friedberg JW, Roschewski MJ, Feldman SA, McIntyre L, Toomey MA, Rosenberg SA. Lymphoma Remissions Caused by Anti-CD19 Chimeric Antigen Receptor T Cells Are Associated With High Serum Interleukin-15 Levels. J Clin Oncol. 2017 Jun 1;35(16):1803-1813. doi: 10.1200/JCO.2016.71.3024. Epub 2017 Mar 14. PMID 28291388
- [Result] Wherry EJ, Kurachi M. Molecular and cellular insights into T cell exhaustion. Nat Rev Immunol. 2015 Aug;15(8):486-99. doi: 10.1038/nri3862. PMID 26205583
- [Result] Oliveira G, Ruggiero E, Stanghellini MT, Cieri N, D'Agostino M, Fronza R, Lulay C, Dionisio F, Mastaglio S, Greco R, Peccatori J, Aiuti A, Ambrosi A, Biasco L, Bondanza A, Lambiase A, Traversari C, Vago L, von Kalle C, Schmidt M, Bordignon C, Ciceri F, Bonini C. Tracking genetically engineered lymphocytes long-term reveals the dynamics of T cell immunological memory. Sci Transl Med. 2015 Dec 9;7(317):317ra198. doi: 10.1126/scitranslmed.aac8265. PMID 26659572
- [Result] Vercellino L, Di Blasi R, Kanoun S, Tessoulin B, Rossi C, D'Aveni-Piney M, Oberic L, Bodet-Milin C, Bories P, Olivier P, Lafon I, Berriolo-Riedinger A, Galli E, Bernard S, Rubio MT, Bossard C, Meignin V, Merlet P, Feugier P, Le Gouill S, Ysebaert L, Casasnovas O, Meignan M, Chevret S, Thieblemont C. Predictive factors of early progression after CAR T-cell therapy in relapsed/refractory diffuse large B-cell lymphoma. Blood Adv. 2020 Nov 24;4(22):5607-5615. doi: 10.1182/bloodadvances.2020003001. PMID 33180899
- [Result] Dean EA, Mhaskar RS, Lu H, Mousa MS, Krivenko GS, Lazaryan A, Bachmeier CA, Chavez JC, Nishihori T, Davila ML, Khimani F, Liu HD, Pinilla-Ibarz J, Shah BD, Jain MD, Balagurunathan Y, Locke FL. High metabolic tumor volume is associated with decreased efficacy of axicabtagene ciloleucel in large B-cell lymphoma. Blood Adv. 2020 Jul 28;4(14):3268-3276. doi: 10.1182/bloodadvances.2020001900. PMID 32702097
- [Result] Casasnovas RO, Ysebaert L, Thieblemont C, Bachy E, Feugier P, Delmer A, Tricot S, Gabarre J, Andre M, Fruchart C, Mounier N, Delarue R, Meignan M, Berriolo-Riedinger A, Bardet S, Emile JF, Jais JP, Haioun C, Tilly H, Morschhauser F. FDG-PET-driven consolidation strategy in diffuse large B-cell lymphoma: final results of a randomized phase 2 study. Blood. 2017 Sep 14;130(11):1315-1326. doi: 10.1182/blood-2017-02-766691. Epub 2017 Jul 12. PMID 28701367
- [Result] Cottereau AS, Nioche C, Dirand AS, Clerc J, Morschhauser F, Casasnovas O, Meignan M, Buvat I. 18F-FDG PET Dissemination Features in Diffuse Large B-Cell Lymphoma Are Predictive of Outcome. J Nucl Med. 2020 Jan;61(1):40-45. doi: 10.2967/jnumed.119.229450. Epub 2019 Jun 14. PMID 31201248
- [Result] Guidetti A, Dodero A, Lorenzoni A, Pizzamiglio S, Argiroffi G, Chiappella A, Bagnoli F, Marasco V, Carniti C, Monfrini C, Seregni E, Pennisi M, Verderio P, Alessi A, Corradini P. Combination of Deauville score and quantitative positron emission tomography parameters as a predictive tool of anti-CD19 chimeric antigen receptor T-cell efficacy. Cancer. 2023 Jan 15;129(2):255-263. doi: 10.1002/cncr.34532. Epub 2022 Nov 17. PMID 36385707
- [Result] Dodero A, Bramanti S, Di Trani M, Pennisi M, Ljevar S, Chiappella A, Massimo M, Guidetti A, Corrado F, Nierychlewska PM, Di Rocco A, Lorenzini D, Daoud R, De Philippis C, Santoro A, Carlo-Stella C, Corradini P. Outcome after chimeric antigen receptor (CAR) T-cell therapy failure in large B-cell lymphomas. Br J Haematol. 2024 Jan;204(1):151-159. doi: 10.1111/bjh.19057. Epub 2023 Sep 10. PMID 37690811
- [Derived] Dodero A, Ceparano G, Casadei B, Angelillo P, Bramanti S, Tisi MC, Ljevar S, Stella F, Chiappella A, Botto B, Cutini I, Zanirato G, Chiusolo P, Barbui AM, Farina M, Di Rocco A, Grillo G, Olivieri J, Krampera M, Ladetto M, Guidetti A, Zinzani PL, Carniti C, Corradini P. Outcomes of CAR T-cell therapy in high-grade B-cell lymphomas compared to DLBCL: a weighted comparison analysis. Blood Adv. 2025 Dec 23;9(24):6491-6501. doi: 10.1182/bloodadvances.2025016117. PMID 40763273
- [Derived] Stella F, Pennisi M, Chiappella A, Casadei B, Bramanti S, Ljevar S, Chiusolo P, Rocco AD, Tisi MC, Angelillo P, Cutini I, Martino M, Barone A, Bonifazi F, Santoro A, Sora F, Novo M, Barbui AM, Russo D, Musso M, Grillo G, Krampera M, Olivieri J, Brunello L, Cavallo F, Massaia M, Arcaini L, Farina L, Zinzani P, Miceli R, Corradini P. Prospective Validation of CAR-HEMATOTOX and a Simplified Version Predict Survival in Patients with Large B-Cell Lymphoma Treated with Anti-CD19 CAR T-Cells: Data from CART-SIE Study. Transplant Cell Ther. 2025 Apr;31(4):240.e1-240.e9. doi: 10.1016/j.jtct.2025.01.888. Epub 2025 Jan 25. PMID 39870308